CLINICAL TRIAL: NCT04622124
Title: A Phase 1, Single-center, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Study to Access the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food-effect of FCN-207 in Healthy Volunteers
Brief Title: A Safety and Tolerability Study of FCN-207 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fochon Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FCN-207-PhⅠ-001
Record Dates: First submitted 2020-10-15; First posted 2020-11-09 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2021-11

CONDITIONS: Hyperuricemia
Keywords: hyperuricemia; single and multiple ascending doses; food effect
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 Single Ascending Dose (SAD) study (Placebo Comparator): The single ascending dose trial set up 7 dose groups of 2.5, 5, 10, 20, 40, 60 and 80 mg. The 2.5 mg dose group was the exploratory part with open label, while the other dose groups were double-blind. 8 subjects were randomly enrolled in each dose group, 6 of whom received FCN-207 tablets and 2 of whom received placebo. This part of the study evaluated the safety, tolerability, and pharmacokinetic and pharmacodynamic studies of single dose FCN-207 tablets in healthy volunteers.
  Interventions: Drug: Placebo
- Part 2 Food-effect study (Experimental): Twelve subjects were enrolled and randomly divided into two groups. The subjects were given FCN-207 tablets after fasting and high-fat diet with double Cross experiment , and feces samples were collected for metabolism/excretion characteristics study.
  Interventions: Dietary Supplement: fasted vs. high-fat meal
- Part 3 Multiple Ascending Dose (MAD) study (Placebo Comparator): A total of 16 subjects were randomly assigned to each dose group for multiple dose study , including 12 who received FCN-207 tablets and 4 who received placebo for a 10-day administration cycle. The dosage of multiple administration was based on the results of single ascending dose study results , and the method of drug administration refers to the results of the food influence test.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Part 1 Single Ascending Dose (SAD) study
Dietary Supplement: fasted vs. high-fat meal
  Arms: Part 2 Food-effect study
Drug: Placebo
  Arms: Part 3 Multiple Ascending Dose (MAD) study

SUMMARY:
This research study is studying an investigational drug called FCN-207 in healthy adult males or females.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, dose-escalations (SAD and MAD) and food effect study of FCN-207:

Part 1 Single Ascending Dose (SAD) study: randomized, double-blind, placebo-controlled.

Part 2 Food-effect study: single-dose, two-treatment (fasted vs. high-fat meal), two-sequence crossover design.

Part 3 Multiple Ascending Dose (MAD) study: randomized, double-blind, placebo-controlled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy subjects who were aged at 18 - 45 years；
2. Weight ≥ 50 kg，Body Mass Index（BMI）＝ Weight（kg）/（Height）2（m2）， BMI at 19 - 28 kg/m2（Including boundary value）；
3. No birth plan during the trial period and within 6 months after completion and are willing to use non-hormonal contraceptive measures;
4. To understand the research procedure and method, voluntarily participate in the experiment and signed the informed consent；

Exclusion Criteria:

1. Blood uric acid < 4 mg/dL（240 μmol/L）or >7 mg/dL（420 μmol/L）；
2. After inquiry and physical examination，subjects who have had cardiovascular, liver, kidney, gastrointestinal respiratory, neurological, mental, immune, blood, endocrine and metabolic diseases, or clinically significant symptoms/signs, or self-report the history of diseases；
3. Physical examination（Height, weight, breathing, pulse, blood pressure, chest and abdominal examinations, etc）or the laboratory indexes [ Blood routine, urine routine, blood biochemistry ( including myocardial enzyme spectrum ), blood amylase and urine amylase, blood coagulation test, infectious disease screening, etc] were abnormal and have clinical significance；12-lead ECG、B-ultrasonography and chest radiograph is abnormal and have clinical significance.
4. Subjects who have had a history of smoking (more than 5 cigarettes per day) and drinking alcohol (more than 15g of alcohol per day for women and more than 25g for men (15g is equivalent to 450ml of beer, 150ml of wine or 50ml of low-alcohol liquor), more than twice a week), and had a history of drug abuse;
5. According to the investigator's judgment, the subject may be allergic to the test drug or any of its ingredients；
6. Subjects with a history of hyperuricemia and/or gout disease, or have received drugs that affect uric acid synthesis, metabolism and excretions within 1month before the screening; A history of kidney stones or B-mode ultrasonography during screening showed kidney stones;
7. Alanine aminotransferase and/or aspartate aminotransferase >1.5 times normal upper limit, and/or total bilirubin>1.5 times normal upper limit；
8. eCRCL ≤ 90mL/min ，Calculation formula：Male（140-AGE）×BW（KG）/（72×SCR），Female（140-AGE）×BW（KG）/（72×SCR）×0.85，SCR unit：μmol/L /dl；
9. Subjects who have had any surgery within 6 months before screening;
10. Subjects who have had participated in blood donation volume is ≥ 400 ml or have received blood transfusion within 3 months before the screening；
11. Subjects who have had participated in a clinical trial of any drug or medical device within 3 months before the screening；
12. Subject who have had any prescription drugs (proton pump inhibitors and antacids, etc.)、counter drugs、Chinese herbal medicines or food supplements that may affect the drug under the test within 1 months before the random;
13. Subjects who have had any acute illness experience of clinical significance as determined by the investigator within 1 months before the screening;
14. Subjects who have had smoked, drank alcohol, drank xanthine or caffeine-containing food and beverages, exercised vigorously, or had other factors affecting drug absorption, distribution, metabolism, and excretion within 2 days before the random；
15. Hepatitis B surface antigen, hepatitis C antibody, HIV antibody, and syphilis antibody is checked positive person;
16. Females during pregnancy or breastfeeding；
17. Subjects who are not suitable for venous blood sampling collection；
18. The investigator judges that the subject has a disease that affects drug absorption, distribution, metabolism and excretion or can reduce compliance（Cardiovascular, liver, kidney, digestive tract, immune, blood, endocrine, metabolic, cancer, psychoneurosis, etc）；subjects may be in a situation or with a condition that, in the opinion of the investigator, would interfere with optimal participation in the study；
19. Subjects who have had a risk factor for TVT or a family history (i.e., parent, sibling, or child) of short QT syndrome, long QT syndrome, unexplained sudden death, drowning, or infant syndrome in their youth (Less than/equal to age 40);
20. Subjects who have had blood potassium, blood magnesium or blood calcium exceeds the normal range；

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
To quantify the occurrence of adverse events (AEs) reported in all subjects who received study drug | Up to week 4
  Incidence of untoward medical occurrences (adverse event = AE) in a participant who received study drug. Adverse events will be evaluated by dosing cohort and recorded according to NCI CTCAEv5 Common Toxicity Criteria
To determine the occurrence of treatment-emergent adverse events (TEAs) | Up to week 4
  Incidence of untoward medical occurrences (adverse event = AE) attributed to study drug in a participant who received study drug. Adverse events will be evaluated and recorded by dosing cohort according to NCI CTCAEv5 Common Toxicity Criteria
To determine the occurrence of treatment-related adverse events meeting the criteria for dose limiting toxicities (DLTs) | Up to week 4
  Incidence of the DLT population will consist all subjects who received the required amount of study drug during the DLT observation period (single ascending doses group：7 days ，multiple ascending doses：21 days) of study treatment . Treatment related AE is any untoward medical occurrence attributed to study drug in a participant that who received study drug. DLTs are adverse events meeting the protocol-specified criteria, evaluated and recorded according to NCI CTCAEv5 Common Toxicity Criteria will use medical terminology based on the Medical Dictionary for Regulatory Activities Terminology (MedDRA).

SECONDARY OUTCOMES:
Pharmacokinetics (AUC: Area under the plasma concentration-time curve) | 2 weeks
Pharmacokinetics (Cmax: Maximum plasma concentration) | 2 weeks
Pharmacokinetics (Tmax: Time to reach the peak plasma concentration) | 2 weeks
Pharmacokinetics (T1/2: Elimination half-life of plasma concentration) | 2 weeks
Pharmacokinetics (CL/F) | 2 weeks
Pharmacokinetics (Vd/F: Distribution volume / Fraction of dose absorbed) | 2 weeks
Pharmacokinetics (λz：Elimination rate constant) | 2 weeks
Pharmacokinetics (DF) | 2 weeks
Pharmacokinetics (RCmax： Cmax accumulation multiple consecutive times) | 2 weeks
Pharmacokinetics (RAUC：AUC accumulation multiple consecutive times) | 2 weeks

OTHER OUTCOMES:
Pharmacokinetics（CFE：Cumulative fecal excretion） | At week1, 2, 3

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university Third Hospital, Beijing, Beijing Municipality, China